CLINICAL TRIAL: NCT00892762
Title: Travoprost APS Versus Xalatan® in Patient Reported Outcomes and Ocular Surface Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-001
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Ocular hypertension; OAG; OH
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost APS (Experimental): Travoprost APS 40 micrograms/ml eye drop solution, 1 drop in the study eye(s), once daily each evening, for 90 days
  Interventions: Drug: Travoprost APS 40 micrograms/ml eye drop solution
- XALATAN (Active Comparator): Latanoprost 50 micrograms/ml eye drop solution, 1 drop in the study eye(s), once daily each evening, for 90 days
  Interventions: Drug: Latanoprost 50 micrograms/ml eye drop solution

INTERVENTIONS:
Drug: Travoprost APS 40 micrograms/ml eye drop solution — non-BAK (benzalkonium chloride) medication
  Arms: Travoprost APS
Drug: Latanoprost 50 micrograms/ml eye drop solution — BAK-preserved medication
  Other Names: XALATAN®
  Arms: XALATAN

SUMMARY:
The purpose of this study is to understand differences in visual function-related patient-reported outcomes between a non-BAK medication (Travoprost APS) and a BAK-preserved medication (XALATAN®) in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component), or ocular hypertension in at least 1 eye.
* Must be willing and able to discontinue use of any topical ocular medication other than the study medication for the duration of the study.
* Must have had Intraocular Pressure (IOP) controlled with mono-therapy using XALATAN® for at least 1 continuous month prior to Visit 1.
* Women of childbearing potential must meet all of the following conditions at Visit 1:

  * They are not breast-feeding.
  * They have a negative urine pregnancy test at Visit 1.
  * They agree to undertake a urine pregnancy test upon entering and exiting the study.
  * They are not planning to become pregnant during the course of the study.
  * They are currently using, and agree to use adequate birth control methods for the duration of the study.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any abnormality preventing reliable applanation tonometry in the study eye(s).
* Presence of any ocular pathology in either eye seen during the slit lamp or fundus exams, that in the opinion of the Investigator may preclude the safe administration of test article or safe participation in this study.
* Dry eye or keratoconjunctivitis sicca (KCS) which has been, or is currently being, treated with the use of punctal plugs, punctal cautery, Restasis®, or topical ocular corticosteroids.
* Patients who have undergone keratorefractive ocular laser procedures, corneal surgery or surgery to the corneal surface, including but not limited to LASIK and PRK, within 6 months prior to Visit 1.
* Patients who have undergone intraocular or extra-ocular surgery, in either eye, within 6 months prior to Visit 1.
* Any history of ocular infections or inflammatory ocular conditions within the past 3 months in either eye.
* Use of any systemic medications on a chronic basis that have not been on a stable dosing regimen for at least 30 days prior to Visit 1.
* Use of ocular medications other than XALATAN® within 7 days of Visit 1.
* Use of corticosteroids within 30 days of Visit 1.
* Use of contact lenses within 30 days of Visit 1. Concomitant use of contact lenses is also excluded for the duration of the study.
* History of intolerance or hypersensitivity to any component of the test articles.
* Participation in an investigational drug or device study within 30 days of entering this study.
* History or evidence of corneal transplant or transplant variant procedures.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean NEI VFQ-25 composite score at the end of the treatment period (Day 90) | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Ph.D., Study Director — Alcon Research